CLINICAL TRIAL: NCT00253539
Title: A Phase II Study of a Selective Estrogen Receptor Modulator (LY353381) vs. Tamoxifen vs. Placebo in Premenopausal Women With and Increased Risk for Breast Cancer
Brief Title: Arzoxifene or Tamoxifen in Preventing Breast Cancer in Premenopausal Women at High Risk for Breast Cancer
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: The Cleveland Clinic (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: G Thomas Budd, MD, Cleveland Clinic Foundation/Taussig Cancer Institute
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: CASE-CCF-4713; P30CA043703 (NIH)
Record Dates: First submitted 2005-11-11; First posted 2005-11-15 (Estimated); Last update posted 2011-04-13 (Estimated); Status verified 2011-04

CONDITIONS: Breast Cancer; Hereditary Breast/Ovarian Cancer (brca1, brca2)
Keywords: hereditary breast/ovarian cancer (BRCA1, BRCA2); breast cancer
MeSH Terms: conditions — Breast Neoplasms; Hereditary Breast and Ovarian Cancer Syndrome | interventions — Tamoxifen

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- Arm I (Experimental): Participants receive oral tamoxifen once daily for 6 months in the absence of disease progression or unacceptable toxicity. After the completion of 6 months of treatment, participants are offered the opportunity to continue treatment for an additional 6 months.
  Interventions: Drug: tamoxifen citrate
- Arm II (Experimental): Participants receive oral arzoxifene once daily for 6 months in the absence of disease progression or unacceptable toxicity. After the completion of 6 months of treatment, participants are offered the opportunity to continue treatment for an additional 6 months.
  Interventions: Drug: arzoxifene hydrochloride
- Arm III (Placebo Comparator): Participants receive an oral placebo once daily once daily for 6 months in the absence of disease progression or unacceptable toxicity. After the completion of 6 months of treatment, participants are offered treatment with arzoxifene for an additional 6 months.
  Interventions: Drug: arzoxifene hydrochloride; Other: placebo

INTERVENTIONS:
Drug: arzoxifene hydrochloride — Given orally
  Arms: Arm II; Arm III
Drug: tamoxifen citrate — Given orally
  Arms: Arm I
Other: placebo — Given orally
  Arms: Arm III

SUMMARY:
RATIONALE: Chemoprevention is the use of certain drugs to keep cancer from forming, growing, or coming back. Estrogen can cause the growth of breast cancer cells. Hormone therapy using arzoxifene or tamoxifen may prevent breast cancer by lowering the amount of estrogen the body makes. The use of arzoxifene or tamoxifen may keep breast cancer from forming in women at high risk for breast cancer.

PURPOSE: This randomized phase II trial is studying arzoxifene to see how well it works compared to tamoxifen or a placebo in preventing breast cancer in premenopausal women at high risk for breast cancer.

DETAILED DESCRIPTION:
OBJECTIVES:

* Compare the effect of arzoxifene vs tamoxifen vs placebo on surrogate endpoints biomarkers, especially systemic insulin-like growth factor levels, in women at high risk for breast cancer.
* Compare the toxic effects, biologic effects, clinical pharmacology, and pharmacodynamics of these drugs in these participants.
* Determine the effect of these drugs on surrogate endpoint biomarkers in participants with BRCA1 and BRCA2 mutations.
* Determine the feasibility of a chemoprevention study in participants with a strong family history of breast cancer.

OUTLINE: This is a randomized, placebo-controlled, double-blind study. Participants are randomized to 1 of 3 treatment arms.

* Arm I: Participants receive oral tamoxifen once daily.
* Arm II: Participants receive oral arzoxifene once daily.
* Arm III: Participants receive an oral placebo once daily. In all arms, treatment continues for 6 months in the absence of disease progression or unacceptable toxicity. After the completion of 6 months of treatment, participants are offered the opportunity to continue treatment with their assigned study drug for an additional 6 months. Participants randomized to receive placebo are offered treatment with arzoxifene for an additional 6 months.

After completion of study treatment, participants are followed annually.

PROJECTED ACCRUAL: A total of 120 participants will be accrued for this study.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Estimated probability of carrying a BRCA1 or BRCA2 mutation ≥ 10% AND meets one of the following criteria:

  * Participants must have first-degree relatives (FDRs)* or second-degree relatives (SDRs)* (with an intervening male relative) with breast or ovarian cancer who satisfy one of the following criteria:

    * High-risk breast/ovarian cancer (non-Jewish families)

      * One FDR ≤ 40 years old** diagnosed with breast cancer
      * At least two FDRs or SDRs diagnosed with breast cancer at ≤ 50 years old OR had bilateral breast cancer
      * One FDR or one SDR diagnosed with breast cancer at ≤ 50 years old OR had bilateral breast cancer AND one FDR or SDR diagnosed with ovarian cancer
      * Three FDRs and/or SDRs diagnosed with breast or ovarian cancer (at least one in case of ovarian cancer)
      * Two FDRs and/or SDRs diagnosed with ovarian cancer
      * One male FDR or SDR diagnosed with breast cancer and one FDR or SDR (male or female) diagnosed with breast or ovarian cancer
    * Moderate-risk breast /ovarian cancer (non-Jewish families)

      * Two FDRs diagnosed with breast cancer with one ≤ 50 years old and/or both < 60 years old
      * One FDR and one SDR (mother or sister and maternal aunt or maternal grandmother) diagnosed with breast cancer if the sum of their ages is ≥ 118 years
      * One FDR and one SDR (mother or sister and paternal aunt or paternal grandmother) diagnosed with breast cancer if the sum of their ages is ≥ 78 years
      * Two SDRs (both maternal or both paternal) diagnosed with breast cancer if the sum of their ages is ≤ 98 years
      * One FDR with ovarian cancer
    * High-risk breast/ovarian cancer (Jewish families )

      * At least one FDR or SDR diagnosed with breast cancer at ≤ 50 years old
      * At least one FDR or SDR diagnosed with ovarian cancer
      * At least one FDR or SDR diagnosed with breast cancer at any age AND one FDR or SDR diagnosed with breast and/or ovarian cancer
      * At least one male FDR or SDR diagnosed with breast cancer NOTE: *FDRs are parents, siblings, and children of the participant; SDRs are aunts, uncles, grandparents, grandchildren, nieces, nephews, or half siblings of the participant

NOTE: **Age is approximated to the earliest age possible (e.g., a relative diagnosed in their 40's should be considered 40)

* Patterns of cancer cases must all be on the maternal or paternal side of the family
* Participants not meeting any of the above FDR or SDR criteria may provide medical documentation stating that they, a FDR, or a SDR carry BRCA1 or BRCA2 mutations

  * Participants with a prior history of breast cancer are eligible provided they have a remaining breast that has not been irradiated, all therapy for breast cancer was completed more than 2 years ago, and they are premenopausal
  * No ovarian cyst during screening
  * No more than 12 months since prior Pap smear with normal cytological results OR human papilloma virus negative if atypical squamous cells of uncertain significance (ASCUS) present
* No higher degrees of atypia beyond ASCUS on Pap smear

  * No known history of osteoporosis (bone mineral density > 1.5 standard deviations below young adult norms)
  * Hormone receptor status
* Not specified

PATIENT CHARACTERISTICS:

Menopausal status

* Premenopausal, as defined by 1 of the following:

  * Last menstrual period < 6 months ago
  * Less than 45 years old AND underwent partial hysterectomy OR follicle-stimulating hormone within institutional pre-menopausal range within the past 3 months

Sex

* Female

Performance status

* ECOG 0-1

Life expectancy

* More than 2 years

Hematopoietic

* WBC ≥ 3,000/mm^3
* Platelet count ≥ 125,000/mm^3
* Hemoglobin ≥ 10 g/dL

Hepatic

* Bilirubin ≤ 1.5 mg/dL
* AST < 2 times upper limit of normal (ULN)
* Albumin ≥ 3.0 g/dL
* PT/PTT ≤ 1.25 times ULN

Renal

* Creatinine ≤ 1.5 mg/dL OR
* Creatinine clearance ≥ 60 mL/min

Cardiovascular

* No history of deep venous thrombosis

Pulmonary

* No history of pulmonary embolism

Other

* Not pregnant or nursing
* Negative pregnancy test
* Fertile participants must use effective barrier-method contraception during and for 3 months after completion of study treatment
* No other malignancy within the past 2 years except curatively treated basal cell or squamous cell skin cancer or cervical cancer ≤ stage I
* No known addiction
* Not undergoing treatment for an illicit drug addiction
* Willing and able to undergo required study procedures (e.g., research-related breast biopsies)

PRIOR CONCURRENT THERAPY:

Chemotherapy

* More than 2 years since prior chemotherapy

Endocrine Therapy

* At least 3 months since prior oral contraceptives or intramuscular progestational agent
* At least 3 months since prior luteinizing-hormone releasing hormone (LHRH) agonists or antagonists if agent was administered daily or monthly
* At least 6 months since prior LHRH agonists or antagonists if agent was administered every 3 months
* At least 6 months since prior antiestrogens (e.g., tamoxifen, toremifene, and raloxifene)
* No concurrent progestational or contraceptive agents

Radiotherapy

* See Disease Characteristics
* More than 2 years since prior radiotherapy

Surgery

* No prior prophylactic bilateral mastectomy

Other

* No concurrent cholestyramine
* No concurrent routine warfarin, bromocriptine, or phenobarbital
* No other concurrent investigational agents

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 3 (Actual)
Dates: Start 2002-01; Primary Completion 2005-04 (Actual); Study Completion 2005-04 (Actual)

PRIMARY OUTCOMES:
Ki67 in breast tissue of enrolled patients
  The primary endpoint was changed in Ki67 in breast tissue of enrolled patients

SECONDARY OUTCOMES:
Toxicity

CONTACTS AND LOCATIONS:
Overall Officials: George T. Budd, MD, Study Chair — The Cleveland Clinic